CLINICAL TRIAL: NCT02396342
Title: A Phase I/II, Open-label, Uncontrolled, Single-dose, Dose-ascending, Multi-centre Trial Investigating an Adeno-associated Viral Vector Containing a Codon-optimized Human Factor IX Gene (AAV5-hFIX) Administered to Adult Patients With Severe or Moderately Severe Hemophilia B
Brief Title: Trial of AAV5-hFIX in Severe or Moderately Severe Hemophilia B
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CT-AMT-060-01
Record Dates: First submitted 2015-03-04; First posted 2015-03-24 (Estimated); Results first posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Hemophilia B
Keywords: Hemophilia B, gene therapy
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): AAV5-hFIX 5 × 10E12 gc/kg intravenous single infusion
  Interventions: Genetic: AAV5-hFIX
- Cohort 2 (Experimental): AAV5-hFIX 2 × 10E13 gc/kg intravenous single infusion
  Interventions: Genetic: AAV5-hFIX

INTERVENTIONS:
Genetic: AAV5-hFIX — AAV5hFIX gene therapy
  Other Names: AAV5 containing a codon-optimized human factor IX gene

SUMMARY:
This study evaluates how safe gene therapy treatment with AAV5-hFIX is in adult patients with severe or moderately severe hemophilia B and severe bleeding type.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age ≥ 18 years
3. Patients with congenital hemophilia B classified as one of the following:

   * Known severe FIX deficiency with plasma FIX activity level < 1% and a severe bleeding phenotype defined by one of the following:

     * Currently on prophylactic FIX replacement therapy for a history of bleeding
     * Currently on on-demand therapy with a current or past history of frequent bleeding defined as four or more bleeding episodes in the last 12 months or chronic hemophilic arthropathy (pain, joint destruction, and loss of range of motion) in one or more joints
   * Known moderately severe FIX deficiency with plasma FIX activity level between ≥ 1% and ≤ 2% and a severe bleeding phenotype defined by one of the following:

     * Currently on prophylactic FIX replacement therapy for a history of bleeding
     * Currently on on-demand therapy with a current or past history of frequent bleeding defined as four or more bleeding episodes in the last 12 months or chronic hemophilic arthropathy (pain, joint destruction, and loss of range of motion) in one or more joints
4. More than 150 previous exposure days of treatment with FIX protein.
5. Acceptance to use a condom during sexual intercourse in the period from Investigational Medicinal Product (IMP) administration until AAV5 has been cleared from semen, as evidenced by the central laboratory from negative analysis results for at least 3 consecutively collected semen samples (this criterion is applicable also for subjects who are surgically sterilized)
6. Following receipt of verbal and written information about the trial, the subject has provided signed informed consent before any trial related activity is carried out.

Exclusion Criteria:

1. History of FIX inhibitors measured to be ≥ 0.6 Bethesda Units (BU)/mL
2. FIX inhibitors ≥ 0.6 BU/mL at Visit 1 (measured by the local laboratory)
3. Neutralizing antibodies against AAV5 at Visit 1 (measured by the central laboratory)
4. Visit 1 laboratory values (measured by the central laboratory):

   * alanine aminotransferase > 2 times upper normal limit
   * aspartate aminotransferase > 2 times upper normal limit
   * total bilirubin > 2 times upper normal limit
   * alkaline phosphatase > 2 times upper normal limit
   * creatinine > 1.5 times upper normal limit
5. Positive HIV serological test at Visit 1, not controlled with anti-viral therapy as shown by cluster of differentiation 4+ counts ≤ 200 per μL or by a viral load of >200 copies per mL (measured by the central laboratory)
6. Active infection with Hepatitis B or C virus as reflected by Hepatitis B Surface Antigen (HBsAg), Hepatitis B extracellular Antigen (HBeAg), Hepatitis B Virus DeoxyriboNucleic Acid (HBV DNA) or Hepatitis C Virus RiboNucleic Acid (HCV RNA) positivity, respectively, at Visit 1 (measured by the central laboratory).
7. History of Hepatitis B or C exposure, currently controlled by antiviral therapy
8. Any coagulation disorder other than hemophilia B
9. Thrombocytopenia, defined as a platelet count below 50 × 10E9 / L, at Visit 1 (measured by the central laboratory)
10. Body mass index < 16 or ≥ 35 kg/m2
11. Planned surgery for the initial 6 months after IMP administration in this trial
12. Previous arterial or venous thrombotic event (e.g. acute myocardial infarction, cerebrovascular disease and venous thrombosis)
13. Active severe infection or any other significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease, alcoholism, drug dependency or any other psychological disorder evaluated by the investigator to interfere with adherence to the protocol procedures or with the degree of tolerance to the IMP
14. Known significant medical condition including disseminated intravascular coagulation, fibrinolysis and liver fibrosis which, in the opinion of the investigator, may confound, contraindicate or limit the interpretation of either safety or efficacy data
15. Known history of an allergic reaction or anaphylaxis to FIX products
16. Known uncontrolled allergic conditions or allergy/hypersensitivity to any component of the IMP excipients
17. Previous gene therapy treatment and/or previous participation in a gene therapy clinical trial
18. Receipt of an experimental agent within 60 days prior to Visit 1
19. Current participation or anticipated participation within one year after IMP administration in this trial in any other interventional clinical trial involving drugs or devices.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: uniQure Clinical Trials, Study Director — UniQure Biopharma B.V.
Locations (7):
- uniQure Investigative Site, Copenhagen, Denmark
- Germany (2):
  - uniQure Investigative Site, Berlin
  - uniQure Investigative Site, Frankfurt
- Netherlands (4):
  - uniQure Investigative Site, Amsterdam
  - uniQure Investigative Site, Groningen
  - uniQure Investigative Site, Rotterdam
  - uniQure Investigative Site, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miesbach W, Meijer K, Coppens M, Kampmann P, Klamroth R, Schutgens R, Tangelder M, Castaman G, Schwable J, Bonig H, Seifried E, Cattaneo F, Meyer C, Leebeek FWG. Gene therapy with adeno-associated virus vector 5-human factor IX in adults with hemophilia B. Blood. 2018 Mar 1;131(9):1022-1031. doi: 10.1182/blood-2017-09-804419. Epub 2017 Dec 15. PMID 29246900

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients with congenital haemophilia B. Known severe FIX deficiency with plasma FIX activity level < 1% and a severe bleeding phenotype.
  Known moderately severe FIX deficiency with plasma FIX activity level between ≥ 1% and ≤ 2% and a severe bleeding phenotype.
  More than 150 previous exposure days of treatment with FIX protein
Groups:
- AAV5-hFIX Low Dose (Cohort 1): AAV5-hFIX 5 × 10E12 gc/kg intravenous single infusion
  AAV5-hFIX: AAV5hFIX gene therapy
- AAV5-hFIX High Dose (Cohort 2): AAV5-hFIX 2 × 10E13 gc/kg intravenous single infusion
  AAV5-hFIX: AAV5hFIX gene therapy
Period: Overall Study
Arm/Group | AAV5-hFIX Low Dose (Cohort 1) | AAV5-hFIX High Dose (Cohort 2)
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set which was comprised of all dosed subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | AAV5-hFIX Low Dose (Cohort 1) | AAV5-hFIX High Dose (Cohort 2) | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (15.9) | 38.2 (5.9) | 49.2 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 3 | 3 | 6
  Denmark | 1 | 0 | 1
  Germany | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: From AMT-060 infusion through end of study (5 years post-dose)
Population: Full Analysis Set (FAS) which was comprised of all dosed subjects
Measure: Number; unit: participants
Arm/Group | AAV5-hFIX Low Dose (Cohort 1) | AAV5-hFIX High Dose (Cohort 2)
Number analyzed (Participants) | 5 | 5
participants | 5 | 5

2. Secondary Outcome: FIX-replacement-therapy-free FIX Activity
Description: FIX activity measured any time from 72 hours after latest FIX replacement therapy administration and until next administration of FIX replacement therapy. Only assessments performed more than 10 days after most recent FIX-replacement therapy administration included.
Time Frame: From AMT-060 infusion through end of study (5 years post-dose)
Population: FAS. Only assessments performed more than 10 days after most recent FIX-replacement therapy administration included.
Measure: Mean (Standard Deviation); unit: Percent FIX activity
Arm/Group | AAV5-hFIX Low Dose (Cohort 1) | AAV5-hFIX High Dose (Cohort 2)
Number analyzed (Participants) | 4 | 5
Percent FIX activity
  one-stage aPTT assay: number analyzed (Participants) | 4 | 4
  one-stage aPTT assay | 7.43 (1.28) | 6.60 (1.96)
  amidolytic/chromogenic assay | 4.58 (2.88) | 4.74 (1.43)

3. Secondary Outcome: Total Annualized Bleeding Rate (ABR)
Description: Annualized: Sum of post-treatment bleeding episodes divided by subjects' average number of years (365.25 days) from treatment start to until the data cutoff date.
Time Frame: From AMT-060 infusion through end of study (5 years post-dose)
Population: FAS. One subject in Cohort 2 did not report any bleeding information for the period 1 year prior to screening. Post-tapering period = from discontinuation of FIX prophylaxis until data cutoff.
Measure: Mean (Standard Deviation); unit: bleeds/year/subject
Arm/Group | AAV5-hFIX Low Dose (Cohort 1) | AAV5-hFIX High Dose (Cohort 2)
Number analyzed (Participants) | 5 | 5
bleeds/year/subject
  One Year Prior to Screening: number analyzed (Participants) | 5 | 4
  One Year Prior to Screening | 14.40 (5.73) | 4.00 (3.16)
  Post-tapering Period | 5.39 (5.94) | 0.71 (0.58)

4. Secondary Outcome: Total Consumption of FIX Replacement Therapy
Time Frame: From AMT-060 infusion through end of study (5 years post dose).
Population: FAS. Post-tapering period = from discontinuation of FIX prophylaxis until data cutoff.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | AAV5-hFIX Low Dose (Cohort 1) | AAV5-hFIX High Dose (Cohort 2)
Number analyzed (Participants) | 5 | 5
IU
  One year prior to screening | 326532 (234900) | 233778 (156873)
  Post-tapering period | 252950 (222790) | 85800 (84482)

5. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Quality of Life (QoL) Scores
Description: Scores range from 0 to 100, with a higher score defining a more favorable health state.
Time Frame: From AMT-060 infusion through the end of study (5 years post dose)
Population: FAS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AAV5-hFIX Low Dose (Cohort 1) | AAV5-hFIX High Dose (Cohort 2)
Number analyzed (Participants) | 5 | 5
score on a scale
  Physical Functioning | 0.00 (10.00) | -7.00 (9.75)
  Role-Physical | -15.00 (8.39) | -10.00 (22.79)
  Bodily Pain | -9.00 (9.00) | 1.20 (14.81)
  General Health | -0.80 (20.22) | -2.40 (8.99)
  Vitality | -11.25 (19.96) | -6.25 (12.50)
  Social Functioning | -20.00 (25.92) | -5.00 (14.25)
  Role-Emotional | -13.33 (27.39) | -10.00 (13.69)
  Mental Health | -13.00 (22.80) | -9.00 (12.94)

6. Secondary Outcome: Time to Vector DNA Stopped Shedding From Blood, Nasal Secretions, Saliva, Urine, Feces, and Semen
Time Frame: From AMT-060 infusion through end of study (5 years post dose).
Population: FAS. Subject in Cohort 1 was unable to produce semen due to a historical medical condition.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AAV5-hFIX Low Dose (Cohort 1) | AAV5-hFIX High Dose (Cohort 2)
Number analyzed (Participants) | 5 | 5
Days
  Blood | 508.8 (261.7) | 705.4 (245.1)
  Nasal secretions | 83.4 (41.7) | 108.4 (66.0)
  Saliva | 75.8 (38.4) | 129.2 (48.9)
  Urine | 46.4 (20.9) | 82.0 (41.1)
  Feces | 74.0 (25.7) | 165.0 (68.9)
  Semen: number analyzed (Participants) | 4 | 5
  Semen | 227.8 (147.7) | 157.2 (78.4)

7. Secondary Outcome: Number of Subjects Developing Neutralizing Antibodies to AAV5
Time Frame: From AMT-060 infusion through end of study (5 years post dose)
Population: FAS
Measure: Number; unit: participants
Arm/Group | AAV5-hFIX Low Dose (Cohort 1) | AAV5-hFIX High Dose (Cohort 2)
Number analyzed (Participants) | 5 | 5
participants | 5 | 5

8. Secondary Outcome: Total IgG and IgM Antibody Titers to AAV5
Description: For subjects with a titer of 109350 and 50, the actual titer is >109350 and <50.
Time Frame: AMT-060 infusion through end of study (5 years post dose)
Population: FAS
Measure: Number; unit: Titer
Arm/Group | AAV5-hFIX Low Dose (Cohort 1) | AAV5-hFIX High Dose (Cohort 2)
Number analyzed (Participants) | 5 | 5
Titer
  IgG (subject 1) | 79499 | 109350
  IgG (subject 2) | 109350 | 109350
  IgG (subject 3) | 109350 | 109350
  IgG (subject 4) | 109350 | 107344
  IgG (subject 5) | 109350 | 109350
  IgM (subject 1) | 56 | 30071
  IgM (subject 2) | 1321 | 20000
  IgM (subject 3) | 557 | 6649
  IgM (subject 4) | 11568 | 50
  IgM (subject 5) | 809 | 50

9. Secondary Outcome: Number of Subjects With a Positive AAV5 Capsid-specific T Cell Response
Description: Specific AAV5 response (results >17 SFC/million PBMCs) were regarded as positive.
Time Frame: From AMT-060 infusion through 26 weeks post-dose
Population: FAS
Measure: Number; unit: participants
Arm/Group | AAV5-hFIX Low Dose (Cohort 1) | AAV5-hFIX High Dose (Cohort 2)
Number analyzed (Participants) | 5 | 5
participants | 1 | 0

10. Secondary Outcome: Number of Subjects With Antibodies to FIX
Time Frame: From AMT-060 infusion through the end of study (5 years post dose)
Population: FAS
Measure: Number; unit: participants
Arm/Group | AAV5-hFIX Low Dose (Cohort 1) | AAV5-hFIX High Dose (Cohort 2)
Number analyzed (Participants) | 5 | 5
participants | 1 | 0

11. Secondary Outcome: Number of Subjects With FIX Inhibitors
Time Frame: From AMT-060 infusion through the end of study (5 years post dose)
Population: FAS
Measure: Number; unit: participants
Arm/Group | AAV5-hFIX Low Dose (Cohort 1) | AAV5-hFIX High Dose (Cohort 2)
Number analyzed (Participants) | 5 | 5
participants | 0 | 0

12. Secondary Outcome: Number of Subjects With Clinically Significant Inflammatory Markers: IL-1β, IL-2, IL-6, INFγ, MCP-1
Time Frame: From AMT-060 infusion through 18 weeks post dose
Population: FAS
Measure: Number; unit: participants
Arm/Group | AAV5-hFIX Low Dose (Cohort 1) | AAV5-hFIX High Dose (Cohort 2)
Number analyzed (Participants) | 5 | 5
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years post-dose
Arm/Group | AAV5-hFIX Low Dose (Cohort 1) | AAV5-hFIX High Dose (Cohort 2)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/5 | 2/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AAV5-hFIX Low Dose (Cohort 1) (N=5) | AAV5-hFIX High Dose (Cohort 2) (N=5)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Renal Colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus Ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AAV5-hFIX Low Dose (Cohort 1) (N=5) | AAV5-hFIX High Dose (Cohort 2) (N=5)
Haematoma (Vascular disorders) | 0 (0) | 1 (2)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Influenza like illness (General disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (2)
Malaise (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Drug ineffective (General disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (5) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (2) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (10) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (2) | 3 (8)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT02396342/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT02396342/SAP_001.pdf